CLINICAL TRIAL: NCT01580033
Title: Immunogenicity and Safety Study of A Group A, C Polysaccharide Meningococcal and Type b Haemophilus Influenzal Conjugate Vaccine in Aged 3-5 Months: A Phase 3 Clinical Trial
Brief Title: Phase 3 Study of A Group A, C Polysaccharide Meningococcal and Type b Haemophilus Influenzal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Royal (Wuxi) Biological Co., LTD (Other)
Responsible Party: Principal Investigator, Fengcai Zhu, Director of Vaccine Clinical Evaluation Center in Jiangsu Province Centers for Disease Control and Prevention, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT009
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Meningitis; Influenza
Keywords: immunogenicity; safety; group A, C polysaccharide meningitis; type b haemophilus Influenza
MeSH Terms: conditions — Meningitis; Influenza, Human | interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A+C+hib Conjugate Vaccine (Experimental): 600 infants aged 3-5 months, will be vaccinated on day0, 28, 56
  Interventions: Biological: A+C+hib Conjugate Vaccine; Biological: Placebo
- Walvax AC vaccine, Pasteur Hib vaccine (Active Comparator): 300 infants aged 3-5 months, will be vaccinated on day0, 28, 56
  Interventions: Biological: A+C Vaccine; Biological: Hib vaccine

INTERVENTIONS:
Biological: A+C+hib Conjugate Vaccine — The group A, C polysaccharide meningococcal and type b haemophilus influenzal conjugate vaccine (Wuxi Royal Biological Co., LTD, 20110101) will be administered on one arm, intramuscularly, per 0.5ml dose
  Arms: A+C+hib Conjugate Vaccine
Biological: Placebo — Placebo will be administered intramuscularly on the other arm, intramuscularly, per 0.5ml dose
  Arms: A+C+hib Conjugate Vaccine
Biological: A+C Vaccine — The group A, C polysaccharide meningococcal vaccine (Yunnan Walvax Biotechnology Co., LTD, 20101202) will be administered intramuscularly on one arm, per 0.5ml dose
  Arms: Walvax AC vaccine, Pasteur Hib vaccine
Biological: Hib vaccine — The type b haemophilus influenzal vaccine (Sanofi Pasteur Limited) will be administered intramuscularly on the other arm, per 0.5ml dose
  Arms: Walvax AC vaccine, Pasteur Hib vaccine

SUMMARY:
Haemophilus influenzae is an important pathogen which can cause primary infection and respiratory viral infection in infants and leaded to secondary infections. The infection of haemophilus is a major cause of morbidity and mortality in infants and children. At present, the developed conjugant Hib vaccine is proved to be safe and effective. Because Hib vaccine can prevent meningitis, pneumonia, epiglottis inflammation and other serious infection caused by Hib bacteria, the WHO suggested that Hib vaccine should be included in the infant's normal immune programming.

Since the use of meningitis aureus polysaccharide vaccine, incidence of a disease in recent years is declined and maintain to the level of 0.5 per 1/100 thousand. But meningitis aureus polysaccharide vaccine with a relatively poor immune response in the infants under the age of two, and the remaining 60% with a low antibody level and a short duration.

The immunogenicity and safety of this vaccine has been proved in older children aged 6-23 months and 2-5 years. And in the phase I study which was conducted in February, 2012, the safety profile of this vaccine is proved to be acceptable in infants aged 3-5 months. The phase III study is aimed to further evaluate the safety and the immunization of the vaccine. The objective of this study is to evaluate the safety of the group A, C polysaccharide meningococcal and type b haemophilus influenzal conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 3 to 5 months, normal intelligence.
* The subjects' guardians are able to understand and sign the informed consent.
* Healthy subjects confirmed by medical history questioning, physical examination and clinical decision and in accordance with vaccination requirements of the investigational vaccine.
* Subjects who can comply with the requirements of the clinical trial program according to the researcher's views.
* Subjects who have never received group A, C polysaccharide meningococcal vaccine and type b haemophilus Influenzal vaccine.
* Subjects with temperature<=37°C on axillary setting.

Exclusion Criteria for the first vaccination:

* Subject who has a medical history of Meningitis;
* Subject who has a medical history of any of the following: allergies, seizures, epilepsy, encephalopathy history and so on;
* Subject who is allergic with tetanus toxoid components;
* Subject suffering from thrombocytopenia or other coagulation disorder may lead to contraindication to intramuscular injection;
* Subject who has a history of allergic reactions;
* Any known immunological dysfunction;
* Had received gamma globulin or immune globulin, in the past two weeks
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of other research medicines in last 1 month
* Any prior administration of attenuated live vaccine in last 28 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Subject suffering from congenital malformations, developmental delay or serious chronic disease;
* Any acute infections
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion Criteria for the second or third vaccination:

* Had any Grade 3 or Grade 4 adverse reactions or events associated with investigational vaccine occurred since the vaccination
* Any situation meets the exclusion criteria for first dose;
* Any condition the investigator believed may affect the evaluation of the vaccine.

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The seroconversion rate of antibody against group A, C polysaccharide meningitis in infants aged 3-5 months | 4 weeks (28±3 days) after the infant series
  the seroconversion rate of antibody against group A, C polysaccharide meningitis in infants aged 3-5 months when measured 4 weeks (28±3 days) after the infant series (three doses, 28 day apart).
The seroconversion rate of antibody against type b haemophilus influenza in infants aged 3-5 months | 4 weeks (28±3 days) after the infant series
  the seroconversion rate of antibody against type b haemophilus Influenza in infants aged 3-5 months when measured 4 weeks (28±3 days) after the infant series (three doses, 28 day apart)

SECONDARY OUTCOMES:
adverse reactions after the first vaccination in infants aged 3-5 months | 7 days after the first vaccination
  adverse reactions of the investigational vaccines in healthy infants aged 3-5 months for 7 days after the first vaccination
adverse reactions after the second vaccination in infants aged 3-5 months | 7 days after the second vaccination
  adverse reactions of the investigational vaccines in healthy infants aged 3-5 months for 7 days after the second vaccination
adverse reactions after the third vaccination in infants aged 3-5 months | 7 days after the third vaccination
  adverse reactions of the investigational vaccines in healthy infants aged 3-5 months for 7 days after the third vaccination
GMT of antibody against group A, C polysaccharide meningitis in infants aged 3-5 months | 4 weeks (28±3 days) after the infant series
  GMT of antibody against group A, C polysaccharide meningitis in infants aged 3-5 months 4 weeks (28±3 days) after the infant series (three doses, 28 day apart)
GMT of antibody against type b haemophilus Influenza in serum in infants aged 3-5 months | 4 weeks (28±3 days) after the infant series
  GMT of antibody against type b haemophilus Influenza in infants aged 3-5 months 4 weeks (28±3 days) after the infant series (three doses, 28 day apart)

CONTACTS AND LOCATIONS:
Locations (1):
- Funing county Center for Disease Control and Prevention, Yancheng, Jiangsu, China